CLINICAL TRIAL: NCT04353674
Title: Novel Extracorporeal Treatment to Modulate Hyperinflammation in COVID-19 Patients
Brief Title: Modulation of Hyperinflammation in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 115785
Record Dates: First submitted 2020-04-07; First posted 2020-04-20 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS
Keywords: cytokine storm; SLEDD
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single centre, prospective, randomized controlled pilot study with approximately 40 patients to be included: 20 in the control group and 20 patients in the L-MOD-SLEDD group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Patients diagnosed with severe COVID-19: Those admitted to the intensive care unit with evidence of severe respiratory distress syndrome will undergo standard of care
  Interventions: Device: Control group
- SLEDD with a L-MOD (Active Comparator): Patients diagnosed with severe COVID-19: Those admitted to the intensive care unit with evidence of severe respiratory distress syndrome will undergo slow low efficiency daily dialysis for approximately 12 hours, 2 days in a row with a leukocyte modulatory device.
  Interventions: Device: SLEDD with a L-MOD

INTERVENTIONS:
Device: Control group — Patients randomized into this group will receive standard of care for COVID-19 infection
  Arms: Control
Device: SLEDD with a L-MOD — Patients randomized to this group will undergo slow low efficiency daily dialysis for approximately 12 hours, 2 days in a row with a leukocyte modulatory device.
  Arms: SLEDD with a L-MOD

SUMMARY:
Current treatment recommendations are based on very limited evidence and reliant on the deployment of pharmacological strategies of doubtful efficacy, high toxicity, and near universal shortages of supply. On a global scale, there is a desperate need for readily available therapeutic options to safely and cost effectively target the hyper-inflammatory state in ICU patients based on management of severe COVID-19 (evidence of acute respiratory distress syndrome). The study team proposes to use slow low-efficiency daily dialysis to provide an extracorporeal circuit to target this cytokine storm using immunomodulation of neutrophils with a novel leucocyte modulatory device (L-MOD) to generate an anti-inflammatory phenotype, but without depletion of circulating factors.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) is a novel virus that was first reported in December 2019 from Wuhan, China. So far, over 8,000,000 cases have been reported around the globe with >400,000 reported deaths overwhelming hospitals and constraining resources. Death is mainly due to severe acute respiratory syndrome (SARS), requiring mechanical ventilation; however, many hospitals do not have sufficient equipment (i.e. ventilators) to meet the requirements. It had been suggested that severe SARS-related injury may have be related to an excessive reaction of the host's immune system, and a dysregulation of pro-inflammatory cytokines called cytokine storm syndrome. This is characterized by a hyper-inflammatory state leading to fulminant multi-organ failure and elevated cytokine levels. There is a critical and imminent need to identify effective treatments to reduce mortality.

The study team proposes to use slow low-efficiency daily dialysis (SLEDD) to provide an extracorporeal circuit to target this cytokine storm using immunomodulation of neutrophils with a novel leukocyte modulatory device (L-MOD) to generate an anti-inflammatory phenotype, without depletion of circulating factors.

This is a single center, prospective, randomized controlled pilot study in the Critical Care Trauma Centre at Victoria Hospital and Critical Care at University Hospital, London, Ontario. Critical Care at University Hospital is comprised of two units, the Medical-Surgical ICU and the Cardiac Surgical Recovery Unit. The study team will randomize patients requiring ICU admission of COVID-19 into one of two groups; either to standard of care for severe COVID-19 infection or in the active treatment group (standard supportive care + treatment with leukocyte modulation (using L-MOD)), on 1:1, basis. They will know what treatment group they are randomized to.

The study team will use block randomization to randomize the patients into one of these two groups. A computer algorithm is used to generate the randomization sequence in blocks of four (two for standard of care and two for active treatment). This is used to make sure that equal numbers of people get allocated to each arm of the study and that the allocation is equal throughout the lifespan of the trial.

Slow low-efficiency daily dialysis will be performed twice, for approximately 12 hours, 2 days in a row. Due to the nature of the intervention, it is not possible to blind neither the patient nor study team members to the treatment group the patient gets randomized to, with the exception of study team members analyzing the data who will be blinded to the patients' treatment group. Additionally, the study uses robust objective measurements that will be unaffected by the patients' awareness of the group they have been randomized to.

Blood work will be collected before each dialysis treatment initiation, at the end of each session, and then on after day 4 and no later than day 7 in the ICU for the patients receiving intervention. Patients receiving standard of care will have blood work done on day 1, day 2, and after day 4 and no later than day 7 of admission. We will also collect a urine sample from all participants before the first dialysis session only and then again at after day 4 and no later than day 7 in the ICU. End of study will be defined as the last patient discharged from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* High clinical suspicion of COVID-19 from the opinion of both infectious disease specialist (s) and the ICU team
* Evidence of acute respiratory distress syndrome requiring admission to the Critical Care Trauma Centre Medical Surgical ICU, or the Cardiac Surgical Recovery Unit
* Vasopressor support

Exclusion Criteria:

* Pregnant
* Unconfirmed COVID-19
* Chronic immune depression
* Contra-indications to regional citrate anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Efficacy of a L-MOD against controls receiving supportive care in ICU. | Through dialysis, on average of 12 hours, two days in a row
  Efficacy will be evaluated by reduction of vasopressor support (converted to norepinephrine dose equivalents) compared to control group.

SECONDARY OUTCOMES:
Mortality | From date of randomization until the date of death from any cause, whichever came first, assessed up to 2 months
  Time to ICU and hospital discharge compared to case-matched controls
Hospital Discharge | From date of randomization until the date of hospital discharge or death from any cause, whichever came first, assessed up to 2 months
  Time to ICU and hospital discharge compared to case-matched controls
Leukocyte Monitoring | Through dialysis, on average of 12 hours, two days in a row and again on day 5 in the ICU
  Over the course of the disease white blood cells will be monitored (i.e. neutrophils, macrophages...)
Sequential Organ Failure Assessment (SOFA) Score | From date of randomization until the date of ICU discharge or death from any cause, whichever came first, assessed up to 1 months
  Evolution of the Sequential Organ Failure Assessment (SOFA) score. The SOFA score ranges from 0 to 24. The higher score means the worst outcome.
Intubation length | From date of randomization until the date of ICU discharge up to 2 months
  intubation length will be recorded (in day)
Markers of Inflammation | Through dialysis, on average of 12 hours, two days in a row and again after day 4 and no later than day 7 in the ICU
  Evolution of hsCRP during dialysis treatment
Leukocytes and Macrophages | Through dialysis, on average of 12 hours, two days in a row and again after day 4 and no later than day 7 in the ICU
  Characterization of activated/desactivated leukocyte and macrophage subsets in the blood
Myocardial damage | From date of randomization until the date of ICU discharge up to 2 months
  Myocardial damage will be assessed by troponin measurement (ng/mL)
Renal recovery | From date of randomization until the date of ICU discharge up to 2 months
  Renal recovery will be assessed by serum creatinin measurement (micromol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD, Principal Investigator — Western University
Locations (2):
- Canada (2):
  - University Hospital, London, Ontario
  - Victoria Hospital - Critical Care Trauma Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Deng Y, Liu W, Liu K, Fang YY, Shang J, Zhou L, Wang K, Leng F, Wei S, Chen L, Liu HG. Clinical characteristics of fatal and recovered cases of coronavirus disease 2019 in Wuhan, China: a retrospective study. Chin Med J (Engl). 2020 Jun 5;133(11):1261-1267. doi: 10.1097/CM9.0000000000000824. PMID 32209890
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Rosenbaum L. Facing Covid-19 in Italy - Ethics, Logistics, and Therapeutics on the Epidemic's Front Line. N Engl J Med. 2020 May 14;382(20):1873-1875. doi: 10.1056/NEJMp2005492. Epub 2020 Mar 18. No abstract available. PMID 32187459
- [Result] Perlman S, Dandekar AA. Immunopathogenesis of coronavirus infections: implications for SARS. Nat Rev Immunol. 2005 Dec;5(12):917-27. doi: 10.1038/nri1732. PMID 16322745
- [Result] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Result] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Result] Perlman S, Netland J. Coronaviruses post-SARS: update on replication and pathogenesis. Nat Rev Microbiol. 2009 Jun;7(6):439-50. doi: 10.1038/nrmicro2147. PMID 19430490
- [Result] Jiang Y, Xu J, Zhou C, Wu Z, Zhong S, Liu J, Luo W, Chen T, Qin Q, Deng P. Characterization of cytokine/chemokine profiles of severe acute respiratory syndrome. Am J Respir Crit Care Med. 2005 Apr 15;171(8):850-7. doi: 10.1164/rccm.200407-857OC. Epub 2005 Jan 18. PMID 15657466
- [Result] Cheung CY, Poon LL, Ng IH, Luk W, Sia SF, Wu MH, Chan KH, Yuen KY, Gordon S, Guan Y, Peiris JS. Cytokine responses in severe acute respiratory syndrome coronavirus-infected macrophages in vitro: possible relevance to pathogenesis. J Virol. 2005 Jun;79(12):7819-26. doi: 10.1128/JVI.79.12.7819-7826.2005. PMID 15919935
- [Result] He L, Ding Y, Zhang Q, Che X, He Y, Shen H, Wang H, Li Z, Zhao L, Geng J, Deng Y, Yang L, Li J, Cai J, Qiu L, Wen K, Xu X, Jiang S. Expression of elevated levels of pro-inflammatory cytokines in SARS-CoV-infected ACE2+ cells in SARS patients: relation to the acute lung injury and pathogenesis of SARS. J Pathol. 2006 Nov;210(3):288-97. doi: 10.1002/path.2067. PMID 17031779
- [Result] Nicholls JM, Poon LL, Lee KC, Ng WF, Lai ST, Leung CY, Chu CM, Hui PK, Mak KL, Lim W, Yan KW, Chan KH, Tsang NC, Guan Y, Yuen KY, Peiris JS. Lung pathology of fatal severe acute respiratory syndrome. Lancet. 2003 May 24;361(9371):1773-8. doi: 10.1016/s0140-6736(03)13413-7. PMID 12781536
- [Result] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: Guidelines on the Management of Critically Ill Adults with Coronavirus Disease 2019 (COVID-19). Crit Care Med. 2020 Jun;48(6):e440-e469. doi: 10.1097/CCM.0000000000004363. PMID 32224769
- [Result] Ding F, Song JH, Jung JY, Lou L, Wang M, Charles L, Westover A, Smith PL, Pino CJ, Buffington DA, Humes HD. A biomimetic membrane device that modulates the excessive inflammatory response to sepsis. PLoS One. 2011 Apr 14;6(4):e18584. doi: 10.1371/journal.pone.0018584. PMID 21533222
- [Result] Ding F, Yevzlin AS, Xu ZY, Zhou Y, Xie QH, Liu JF, Zheng Y, DaSilva JR, Humes HD. The effects of a novel therapeutic device on acute kidney injury outcomes in the intensive care unit: a pilot study. ASAIO J. 2011 Sep-Oct;57(5):426-32. doi: 10.1097/MAT.0b013e31820a1494. PMID 21317636
- [Result] Humes HD, Sobota JT, Ding F, Song JH; RAD Investigator Group. A selective cytopheretic inhibitory device to treat the immunological dysregulation of acute and chronic renal failure. Blood Purif. 2010;29(2):183-90. doi: 10.1159/000245645. Epub 2010 Jan 8. PMID 20093825
- [Result] Tumlin JA, Galphin CM, Tolwani AJ, Chan MR, Vijayan A, Finkel K, Szamosfalvi B, Dev D, DaSilva JR, Astor BC, Yevzlin AS, Humes HD; SCD Investigator Group. A Multi-Center, Randomized, Controlled, Pivotal Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device in Patients with Acute Kidney Injury. PLoS One. 2015 Aug 5;10(8):e0132482. doi: 10.1371/journal.pone.0132482. eCollection 2015. PMID 26244978